CLINICAL TRIAL: NCT01539070
Title: Design and Feasibility of a Clinical-based Intervention to Prevent Obesity in Preschool Children
Brief Title: Intervention for the Prevention of Obesity in Preschool
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Hospital Infantil de Mexico Federico Gomez (Other); Harvard Pilgrim Health Care (Other); Fogarty International Center of the National Institute of Health (NIH); Inter-American Development Bank (Other); Instituto Nacional de Salud Publica, Mexico (Other); University of Guelph (Other)
Responsible Party: Principal Investigator, Gloria Oliva Martinez Andrade, Investigador Asociado A, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-785-120; HIM/2010/025 (Other Grant/Funding Number: Hospital Infantil de México); 1R03TW008708 (NIH)
Record Dates: First submitted 2012-02-14; First posted 2012-02-27 (Estimated); Results first posted 2014-04-22 (Estimated); Last update posted 2014-04-22 (Estimated); Status verified 2014-03

CONDITIONS: Childhood Obesity
Keywords: Nutritional intervention; Childhood obesity; Physical activity; Feeding practices
MeSH Terms: conditions — Pediatric Obesity; Motor Activity | interventions — Eating

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eating and physical activity counseling (Experimental): Participants randomized to intervention received a 6 week curriculum focused on obesity awareness and prevention. A trained nutritionist led diet, healthy growth and physical activity workshops, while a health educator led workshops on instilling healthy habits and routines in childhood. The nurse provided child care and developed relevant games and activities for children while parents attended the workshops.
  Interventions: Behavioral: Eating and physical activity counseling
- Usual care (No Intervention): According to the existing clinical practice guide within IMSS, obese children may be referred to a nutritionist if the physician considers it necessary, given general dietary advice by the attending physician, or, if necessary, sent for laboratory analyses of blood lipids and glucose. We gave the parents the height and weight results from the measurement of their child and recommended they share results with their physician in their next medical consultation.

INTERVENTIONS:
Behavioral: Eating and physical activity counseling — The parents of overweight children will be invited to attend a total of 6 group sessions (the group will be comprised of 6 children with their parents) on a weekly basis, in which 5 aspects will be dealt with 1) Dietary culture, risk-benefit practices, 2) The process of feeding (acquisition/preparation/service Eating behaviors), 3) Physical activity habits, 4) Importance of weighing/measuring oneself and its meaning, 5) feedback and evaluations. These aspects and contents will be distributed throughout the 6 sessions.
  There will be two more individual session, at 3 and 6 months respectively, for the reinforcement of recommendations provided for the modification of dietary behaviors and physical activity.
  Other Names: Nutritional intervention
  Arms: Eating and physical activity counseling

SUMMARY:
The purpose of this study is to develop, implement and evaluate an intervention focused to change feeding practices and patterns of physical activity of preschool children through providing motivational counseling to the mother. The aim is to prevent obesity in children aged 2 to 4 years 11 months with risk of overweight or with overweight.

DETAILED DESCRIPTION:
Obesity has a multi-causal origin in which participate, in a similar way, the individual behavior and family and community contexts and the social environment.

Participation of primary care services is key to solve the problem. These services have the possibility to detect timely children with high body mass index, and to promote behavior to improve feeding practices and physical activity in both, the child and his family.

The study is divided in two stages:

1. Design of the intervention. The researchers will use qualitative methods to evaluate feeding practices, physical activity and the environment in which such behaviors are generated. In a similar way the care provided by health professionals to overweight and obese children it will be evaluated; this includes the perception that health providers have about this problem. The information will allow identifying risk behavior and healthy behavior, facilitators and obstacles to receive care. The results will serve to define the contents of the intervention.
2. Intervention: The study will take place in four family medicine clinics belonging to the Mexican Institute of Social Security. Two clinics will receive the intervention and two will serve as control. In each clinic, fifty children and their mothers will be recruited. At the intervention clinics, the group of mothers will participate in seven weekly sessions and in two individual sessions at 3 and 6 months after the group sessions finish. During the sessions, the researchers will motivate the mothers to change feeding practices and encourage physical exercise of the children and family, this will improve the chance for their children for healthy growing. The control group will receive the usual care that consists only in the recommendations that the family doctor provides.

The evaluation of the study comprise feasibility and acceptability of the intervention and its effect in the behavior of the mothers in terms of changing feeding practices and practicing physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Children between 2 and 4 years and 11 months of age at the beginning of the study.
* Overweight children, defined as a BMI score of z > = 1.5 and < +3 based on the WHO standards.
* The children's parents accept participation in the study.

Exclusion Criteria:

* Families who plan on changing their address during the study.
* Families whose doctor considers them to be inappropriate for participation in the intervention, as with emotional or mental alterations.
* Children who require a special diet for medical reasons or children with limited motor functioning.

Ages: 24 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 306 (Actual)
Dates: Start 2012-03; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Martínez Andrade, Master, Principal Investigator — Instituto Mexicano del Seguro Social; Ricardo Pérez Cuevas, Doctor, Study Director — Inter-American Development Bank; Elsie Taveras, Doctor, Study Director — Harvard Pilgrim Health Care; Matt Gillman, Doctor, Study Chair — Harvard Pilgrim Health Care
Locations (1):
- Epidemiology and Health Services Research Unit, Coordination of Health Research. Mexican Institute of Social Security, Mexico, D.F., Mexico City, Mexico City, Mexico

REFERENCES:
- [Derived] Martinez-Andrade GO, Cespedes EM, Rifas-Shiman SL, Romero-Quechol G, Gonzalez-Unzaga MA, Benitez-Trejo MA, Flores-Huerta S, Horan C, Haines J, Taveras EM, Perez-Cuevas R, Gillman MW. Feasibility and impact of Creciendo Sanos, a clinic-based pilot intervention to prevent obesity among preschool children in Mexico City. BMC Pediatr. 2014 Mar 20;14:77. doi: 10.1186/1471-2431-14-77. PMID 24649831

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study staff screened 3095 children from March, 2012 to October, 2012 in Mexican Institute of Social Security (IMSS) clinics (Intervention (Ix) n=2111; Usual Care (UC) n=984). Staff approached parents and caregivers in the waiting rooms of clinics, weighed and measured children and parents completed a baseline questionnaire to determine eligibility.
Pre-assignment Details: Of the 3095 (Ix n=2111; UC n=984) children initially screened, 1406 (Ix n=984; UC n=422) were eligible to participate and 306 (Ix n=168; UC n=138) agreed to participate. Of these 306, 189 (Ix n=93; UC n=96 control) participated in both the 3 and 6 month follow-up.
Period: Overall Study
Arm/Group | Eating and Physical Activity Counseling | Usual Care
Started | 168 | 138
Completed | 109 | 99
Not Completed | 59 | 39

BASELINE CHARACTERISTICS:
Groups:
- Eating and Physical Activity Counseling: Eating and physical activity counseling : The parents of overweight children will be invited to attend a total of 6 group sessions (the group will be comprised of 6 children with their parents) on a weekly basis, in which 5 aspects will be dealt with 1) Dietary culture, risk-benefit practices, 2) The process of feeding (acquisition/preparation/service Eating behaviors), 3) Physical activity habits, 4) Importance of weighing/measuring oneself and its meaning, 5) feedback and evaluations. These aspects and contents will be distributed throughout the 6 sessions.
  There will be two more individual session, at 3 and 6 months respectively, for the reinforcement of recommendations provided for the modification of dietary behaviors and physical activity.
- Total: Total of all reporting groups
Arm/Group | Eating and Physical Activity Counseling | Usual Care | Total
Number analyzed (Participants) | 168 | 138 | 306
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 168 | 138 | 306
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 3.34 (0.84) | 3.42 (0.82) | 3.38 (0.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 81 | 64 | 145
  Male | 87 | 74 | 161
Region of Enrollment [Number; unit: participants]
  Mexico | 168 | 138 | 306

OUTCOME MEASURES:

1. Primary Outcome: Change in Children´s Consumption of Foods From Baseline to 3 Months by Intervention Assignment
Description: We asked parents about the average number of servings in the week or month the child consumed each food. We constructed grouped diet variables corresponding to food categories : sweet snacks (sugar-sweetened dairy, sugary cereal, cookies, sweet bread, cake, packaged pastries ], caramel pops, candies and chocolates); fast food (hamburgers, pizza, hot dogs, quesadillas, fried tacos, French fries); savory snacks (packaged snack foods, corn or potato chips); fruit (orange, mango, papaya, watermelon, grapes, apple, banana); vegetables (chard, broccoli, jitomate [tomato], nopales [cactus], chayote [squash], spinach, lettuce, zucchini, carrot); sugar-sweetened beverages (soda, flavored milk, homemade [agua fresca] and packaged fruit drinks); and added sugar in beverages (teaspoons sugar or sweet flavoring added to milk, coffee, tea, or fruit juice).
Time Frame: 0, 3 months
Population: Intent-to-treat analyses with multiple imputation to account for missing data. Were included in the analysis of children between 0 and 3 BMI z score, age between 24 and 59 months and parents signed letter of consent to participate in the study
Measure: Mean (Standard Error); unit: servings/week
Arm/Group | Eating and Physical Activity Counseling | Usual Care
Number analyzed (Participants) | 168 | 138
servings/week
  Vegetables | -0.8 (0.2) | -5.5 (0.2)
  Fruit | 0.1 (0.2) | -1.9 (0.4)
  Water | -0.6 (0.2) | -3.5 (0.2)
  Sweet snacks | -9.7 (0.2) | -6.4 (0.3)
  Fast food | -0.4 (0.0) | -0.2 (0.0)
  Savory snacks | -0.7 (0) | -0.5 (0)
  Sugar-sweetened beverages | -6.0 (0.2) | -3.2 (0.2)
  Added sugar in beverages | -4.0 (0.2) | -1.7 (0.2)
Statistical Analysis 1: Comparison: Eating and Physical Activity Counseling vs Usual Care; In intent-to-treat analyses, we used unadjusted and adjusted multivariate regression models, to examine differences from baseline to 3 months between the intervention and usual care groups. For continuous outcomes, we used linear regression models, and for dichotomous outcomes, we used logistic regression models. To account for clustering by practices, we performed generalized linear mixed models. The Estimator (Est) and Confidence Interval 95% (95% CI)are reported; Test type: Superiority or Other; p < 0.05, Regression, Linear; All Regression models adjusted for clustering by clinic, child age, change in age, BMI z-score, maternal education and occupation, and season; Mean Difference (Final Values) = 6.3, 95% CI 2-sided [1.8 to 10.8] — The change in the average vegetable consumption from baseline to 3 months, the intervention group compared with the usual care group
Statistical Analysis 2: Comparison: Eating and Physical Activity Counseling vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Linear; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-13.6 to 10.3] — The change in the average fruit consumption from baseline to 3 months, the intervention group compared with the usual care group
Statistical Analysis 3: Comparison: Eating and Physical Activity Counseling vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 0.6, 95% CI 2-sided [-5.4 to 6.5] — The change in the average water consumption from baseline to 3 months, the intervention group compared with the usual care group
Statistical Analysis 4: Comparison: Eating and Physical Activity Counseling vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Linear; Mean Difference (Final Values) = -3.9, 95% CI 2-sided [-8.9 to 1.1] — The change in the average sweet snacks consumption from baseline to 3 months, the intervention group compared with the usual care group
Statistical Analysis 5: Comparison: Eating and Physical Activity Counseling vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 0.3, 95% CI 2-sided [-0.5 to 1.1] — The change in the average fast food consumption from baseline to 3 months, the intervention group compared with the usual care group
Statistical Analysis 6: Comparison: Eating and Physical Activity Counseling vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Linear; Mean Difference (Final Values) = -0.3, 95% CI 2-sided [-0.5 to 0.0] — The change in the average savory snacks consumption from baseline to 3 months, the intervention group compared with the usual care group
Statistical Analysis 7: Comparison: Eating and Physical Activity Counseling vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Linear; Mean Difference (Final Values) = -0.7, 95% CI 2-sided [-4.9 to 3.4] — The change in the average sugar-sweetened beverage consumption from baseline to 3 months, the intervention group compared with the usual care group
Statistical Analysis 8: Comparison: Eating and Physical Activity Counseling vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Linear; Mean Difference (Final Values) = -2.2, 95% CI 2-sided [-8.4 to 4.1] — The change in the average added sugar in beverage consumption from baseline to 3 months, the intervention group compared with the usual care group

2. Primary Outcome: Change in Children´s Time of Physical Activity From Baseline to 3 Months by Intervention Assignment
Description: Staff assisted parents in reporting the average time the participating child spent in pre-specified active and sedentary activities during the week and on weekends. For each of the pre-specified activities parents reported time spent in open-ended response format. From these responses we derived total hours/week of physical activity composed of active play (e.g. running, jumping, walking, playing ball, playing in the park, biking, swimming, dancing), as well as total hours/week of screen time, composed of television, DVD/video, and video and computer games.
Time Frame: 0, 3 months
Population: In intent-to-treat analyses, we used unadjusted and adjusted multivariate regression models, to examine differences from baseline to 3 and to 6 months between the intervention and usual care groups.
Measure: Mean (Standard Deviation); unit: hours/week
Arm/Group | Eating and Physical Activity Counseling | Usual Care
Number analyzed (Participants) | 168 | 138
hours/week
  Physical activiy | 2.9 (0.2) | 9.5 (0.4)
  Sleep time | -0.3 (0.0) | -0.1 (0.0)
  Screen time | -2.76 (0.1) | -1.97 (0.1)
Statistical Analysis 1: Comparison: Eating and Physical Activity Counseling vs Usual Care; In intent-to-treat analyses, we used unadjusted and adjusted multivariate regression models, to examine differences from baseline to 3 months between the intervention and usual care groups. For continuous outcomes, we used linear regression models, and for dichotomous outcomes, we used logistic regression models. To account for clustering by practices, we performed generalized linear mixed models. The Estimator (Est) and Confidence Interval 95% (95% CI) are reported; Test type: Superiority or Other; p < 0.05, Regression, Linear; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -11.8, 95% CI 2-sided [-29.1 to 5.5] — The change in mean physical activity between the baseline measurement and 3 months, the intervention group compared with the control group
Statistical Analysis 2: Comparison: Eating and Physical Activity Counseling vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-0.2 to 0.5] — The change in mean sleep time between the baseline measurement and 3 months, the intervention group compared with the control group
Statistical Analysis 3: Comparison: Eating and Physical Activity Counseling; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Linear; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-4.4 to 1.1] — The change in mean screen time between the baseline measurement and 3 months, the intervention group compared with the control group

3. Secondary Outcome: Number of Families That Completed 3 Month Follow-up in Intervention Group and Usual Care Group
Description: We assessed the compliance with the study through attendiance appointments for assessing diet and physical activity.
Time Frame: 3 months
Measure: Number; unit: participants
Arm/Group | Eating and Physical Activity Counseling | Usual Care
Number analyzed (Participants) | 168 | 138
participants | 99 | 99

4. Primary Outcome: Change in Score z of Body Mass Index From Baseline to 3 Months by Intervention Assignment
Description: In order to calculate children's BMI and age and sex specific BMI z-scores at baseline and 3 month follow-up, study staff assessed child's height in meters and weight in kilograms. BMI was calculated as weight in kilograms divided by the square of height in meters.
Time Frame: 0, 3 month
Measure: Mean (Standard Error); unit: z score
Arm/Group | Eating and Physical Activity Counseling | Usual Care
Number analyzed (Participants) | 168 | 138
z score | -0.26 (0.01) | -0.44 (0.01)
Statistical Analysis 1: Comparison: Eating and Physical Activity Counseling vs Usual Care; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Regression, Linear; Mean Difference (Final Values) = 0.15, 95% CI 2-sided [-0.04 to 0.35]

ADVERSE EVENTS:
Description: An educational intervention was performed and did not evaluate adverse effects
Arm/Group | Eating and Physical Activity Counseling | Usual Care
Serious Adverse Events (participants affected / at risk) | 0/168 | 0/138
Other Adverse Events (participants affected / at risk) | 0/168 | 0/138

LIMITATIONS AND CAVEATS:
35% of families did not complete follow-up at 3 months, our primary endpoint. To address the resulting bias from missing data we performed multiple imputation of missing information on covariates and behavioral and BMI outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No